CLINICAL TRIAL: NCT02964442
Title: Brown Adipose Tissue Activation and Energy Expenditure by Capsinoids Stimulation With Trimodality Imaging Using 18-FDG-PET, Fat Fraction MRI and Infrared Thermography
Acronym: TACTICAL-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Institute of Bioengineering and Bioimaging (IBB) (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015/00715
Record Dates: First submitted 2016-11-04; First posted 2016-11-16 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Brown Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsinoids (Experimental): 8 gel capsules equivalent to 12mg
  Interventions: Other: Capsinoids
- Cooling Vest (Experimental): Using Cooling vest (at approxiamately14 degrees Celsius) to cool the body.
  Interventions: Other: Cold Stimulus

INTERVENTIONS:
Other: Capsinoids — 12 mg of Gel capsules
  Arms: Capsinoids
Other: Cold Stimulus — Cooling vest maintain at 14 degree Celsius
  Arms: Cooling Vest

SUMMARY:
Brown adipose tissue (BAT) thermogenesis can be assessed by IR thermography, the accompanying increase metabolic rate can be measured by whole body calorimetry and BAT volume can be precisely measured by MRI. The aim of the study is to validate IRT for BAT thermogenesis against the present gold standard 18-FDG-PET scan, quantify BAT volume by fat fraction MRI and measure the accompanying increase in BMR by whole body calorimetry among healthy euthyroid subjects.

DETAILED DESCRIPTION:
It is now known that human adults do possess viable brown fat in quantities that may be critical for maintenance of a normal basal metabolic rate (BMR) and body weight, dispelling the myth that BAT is only present during infancy for thermoregulation. There are data suggesting that obesity is associated with insufficient BAT. So far the only known and arguably 'gold standard' methodology of BAT imaging in humans is 18-FDG-PET. Yet 18-FDG-PET imaging has significant limitations, given its restricted spatial resolution and its non-trivial level of ionizing radiation (2.8 mSv). The International Commission for Radiological Protection recommends that the radiation exposure for the general public should not exceed 1mSv/year and 1.5 mSv/year from background radiation. In addition, 18-FDG-PET depends on glucose uptake by BAT that does not directly measure its key metabolic activity, namely fatty acid oxidation. Finally, PET scans are very costly. This makes the present gold standard far from ideal as a research tool for investigating BAT physiology. Thus the first objective of this project is to develop an alternative activated BAT imaging method that is not based on ionizing radiation. We are interested in advancing infrared (IR) thermography as a method to assess BAT activity by developing a novel image processing algorithms for IR thermography. Much extant literature describes the use of "average temperature" instead of IR heat flux using the physical principles of radiative heat transfer and thermodynamics to quantify heat from BAT. Also,IR digital still-shots were mostly employed in the past whereas none have reported the analysis of IR flux using a video sequence which more accurately integrates time-varying heat energy output. Without precision in capturing and processing the rich IR data, the value of IR thermography as a tool for BAT research is limited. It is thus crucial to convert the IR images into a readout that reflects energy output. We will thus develop, validate and apply automatic IR image processing with computer software that can efficiently calculate BAT activation. In this proposal we will also improve and validate anatomical fat fraction MRI as a tool for evaluating BAT volumes based on the higher water content in BAT compared with that in WAT. Fat fraction imaging by MRI has been proposed but no proper validation has been done due to the difficulty in matching PET and MRI data on BAT. Instead of using pharmacologic agents (e.g. beta 3-adrenergic receptor agonists such as mirabegron) that can be administered to activate BAT instead of cold stimulus, we will employ capsiate (i.e. capsinoids - non-spicy analogues of capsaicin in peppers and chilies) that have been proven to effectively stimulate BAT in thermoneutral conditions as confirmed by PET scans. We have conducted a preliminary study approved by the DSRB that showed the effectiveness of capsinoids in stimulating BAT. There are publications documenting the use of MRI in distinguishing BAT from WAT, each with their advantages and disadvantages. In this present study, we will perform a proof-of-concept study by simultaneous acquisition of MRI and 18-FDG-PET in a dual-modality fusion MRI-PET scanner available at the Clinical Imaging Research Centre (CIRC) to image BAT in humans, and correlate this with IR thermography of the cervical and supraclavicular regions (SCR) and with metabolic rate accurately measured in a whole body calorimeter. Whole body calorimetry is the real gold standard to assess BAT activity by measuring nonshivering thermogenesis. IR has so far been validated against 18-FDG-PET in mice and rodents, but equivalent validation in humans has not been published. If IR thermography is shown to be equivalent or superior to 18-FDG-PET imaging, it will set a new gold standard in BAT imaging which will be a boon for study of BAT biology in humans.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy with no past history of chronic illnesses
* Aged 21-40 years old Male and female gender
* BMI from 18.5 to 29.9 kg/m2 inclusive
* No prior history of thyroid disease.
* Euthyroid biochemically with FT4 and TSH in the normal ranges

Exclusion Criteria:

* Recent changes in weight of >5% over the past 6 months.
* Attempts to lose weight over the past 6 months.
* Significant changes in diet over the past 6 months.
* Any use of weight reducing drugs in the past 6 months.
* Previous weight reducing surgery.
* Any use of investigational drugs in the past 6 months.
* Subclinical thyroid dysfunction based on thyroid function test.
* Chronic illnesses such as diabetes mellitus or cancer.
* You have a known history of thyroid, liver or kidney disease.
* Use of any prescription medication that cannot be safely discontinued within 14 days prior to study entry.
* Female subjects who are pregnant.
* Oral medications affecting brown fat activity (eg. alpha agonists or blockers, beta agonists or blockers, sympatholytic agents) which the researchers will clarify with you.
* Chronic topical ointment with menthol or capsaicin or use of nasal decongestants.
* History of surgery with metallic clips, staples or stents.
* Presence of cardiac pacemaker or other foreign body in any part of the body.
* History of claustrophobia particularly in a MRI scanner.
* Had a PET scan done within the past 4 months.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Brown adipose tissue activation detection by Imaging using 18-FDG-PET/ MRI. | post consumption of capsinoids capsules for 2 hours
Energy Expenditure using Whole Body Calorimeter. | post consumption of capsinoids capsules for 2 hours
Brown adipose tissue activation detection by Imaging using Infrared Thermography. | post consumption of capsinoids capsules for 2 hours

SECONDARY OUTCOMES:
Brown adipose tissue activation detection by Imaging using 18-FDG-PET/ MRI. | post cold stimulus up to 2 hours
Energy Expenditure using Whole Body Calorimeter. | To measure cold stimulus for 2 hours
Brown adipose tissue activation detection by Imaging using Infrared Thermography. | post cold stimulus up to 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun L, Yan J, Goh HJ, Govindharajulu P, Verma S, Michael N, Sadananthan SA, Henry CJ, Velan SS, Leow MK. Fibroblast Growth Factor-21, Leptin, and Adiponectin Responses to Acute Cold-Induced Brown Adipose Tissue Activation. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e520-31. doi: 10.1210/clinem/dgaa005. PMID 31912874
- [Derived] Sun L, Verma S, Michael N, Chan SP, Yan J, Sadananthan SA, Camps SG, Goh HJ, Govindharajulu P, Totman J, Townsend D, Goh JP, Sun L, Boehm BO, Lim SC, Sze SK, Henry CJ, Hu HH, Velan SS, Leow MK. Brown Adipose Tissue: Multimodality Evaluation by PET, MRI, Infrared Thermography, and Whole-Body Calorimetry (TACTICAL-II). Obesity (Silver Spring). 2019 Sep;27(9):1434-1442. doi: 10.1002/oby.22560. Epub 2019 Jul 13. PMID 31301122
- [Derived] Sun L, Camps SG, Goh HJ, Govindharajulu P, Schaefferkoetter JD, Townsend DW, Verma SK, Velan SS, Sun L, Sze SK, Lim SC, Boehm BO, Henry CJ, Leow MK. Capsinoids activate brown adipose tissue (BAT) with increased energy expenditure associated with subthreshold 18-fluorine fluorodeoxyglucose uptake in BAT-positive humans confirmed by positron emission tomography scan. Am J Clin Nutr. 2018 Jan 1;107(1):62-70. doi: 10.1093/ajcn/nqx025. PMID 29381803